CLINICAL TRIAL: NCT05750134
Title: Endoscopic Sleeve Gastroplasty for Overweight or Moderately Obese Patients: Identification of Predictive Factors for Weight Loss
Brief Title: Endoscopic Sleeve Gastroplasty for Moderate Obesity
Acronym: PLICATURE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); INSERM U996 (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP230192
Record Dates: First submitted 2022-12-07; First posted 2023-03-01 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Obesity
Keywords: Obesity; Endoscopic sleeve gastroplasty; Weight loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Moderately obese patients: Moderately obese patients undergoing endoscopic sleeve gastroplasty
  Interventions: Other: OBPLUS Clinical Database : data analysis; Other: Biological collection "Liver, bile ducts and pancreas": sample analysis

INTERVENTIONS:
Other: OBPLUS Clinical Database : data analysis — The data processed relates to patients cared for in the Hepato-gastroenterology and nutrition department of the Antoine Béclère Hospital at the Assistance Publique - Hôpitaux de Paris (AP-HP. All of the clinical and paraclinical data are collected during the visits and entered into the OBPLUS database (database registered in the AP-HP register). These data will be analyzed in order to identify the predictive factors of the effectiveness of the fundo-plication.
Other: Biological collection "Liver, bile ducts and pancreas": sample analysis — The samples (plasma, serum, saliva, stool) collected during the samples taken as part of the patient's care were the subject of a biological collection "Liver, bile ducts and pancreas". These samples will be analyzed in order to identify the predictive factors of the effectiveness of the fundo-plication.

SUMMARY:
Weight loss is of paramount importance to ameliorate obesity-related complications. Endoscopic sleeve gastroplasty is a new therapeutic option to obtain significant weight reduction in obese patients. Nevertheless, a only a part of patients experience sufficient weight loss to improve comorbidities. A better understanding of mechanisms driving body weight trajectory after endoscopic sleeve gastroplasty may help patient selection and improve efficacy. The main aim of this study is to identify factors associated with weight reduction after endoscopic sleeve gastroplasty in patients with overweight or morbid obesity without indication to bariatric surgery. For this purpose, the investigators conduct a retro-prospective cohort study including patients with overweight or moderate obesity undergoing endoscopic sleeve gastroplasty between March 2017 and March 2023

DETAILED DESCRIPTION:
The prevalence of obesity is increasing worldwide, and it is estimated that one quarter of the world's population will be overweight or obese by 2045. Obesity can lead to complications, including cardiovascular damage (myocardial ischemia and stroke), liver damage (non-alcoholic steatohepatitis and liver cancer), diabetes and extra-hepatic cancers. In this context, achievement of a significant long-term weight loss is of paramount importance to ameliorate patient outcome. Bariatric surgery is the most effective treatment for severe obesity and results in a significant long-term weight loss. However, bariatric surgery is restricted to patients with a BMI >40 kg/m2 or >35 kg/m2 with commodities (hypertension, diabetes, sleep apnoea, NASH). Therefore, the majority of obese patients do not benefit from this procedure. Recent advances in flexible endoluminal endoscopy now provide the tools for transoral endoscopic gastric volume reduction (ESG, endoscopic sleeve gastroplasty). The gastric body is reduced by an endoscopic procedure involving suture plications. This minimally invasive method may be a good therapeutic option to obtain a significant weight reduction in patients with moderate obesity or those with severe obesity and no indication for bariatric surgery (BMI between 35 and 40 kg/m2 without commodities). In this context this study aims to identify predictive factors of weight loss following ESG and explore changes of metabolic parameters, metabolomic profiles and gut microbiota profiles. This is a retro-prospective cohort study including patients with moderate obesity undergoing ECG between March 2017 and September 2023. Clinical parameters (weight, high, BMI, weight fluctuations), serum metabolic parameters (standard lipid profile, lipoprotein levels, fasting plasma glucose, insulin levels, C-peptide levels, hemoglobin A1c) and liver function test parameters (standard biology, transient elastometry, Fibrotest®, Actitest®, abdominal ultrasound) are systematically collected for all patients before ESG and then at three- and twelve-month post-ESG. Samples of serum, plasma, stools and saliva are also systematically collected for research purpose before ESG and then at three- and twelve-month post-ESG. Each sample is stored at -80°C for subsequent analysis. Metabolomic/lipidomic analysis will be used to quantify metabolite and lipid species in serum/plasma samples. Metagenomic analysis will be used to characterise faecal and salivary microbiota profiles.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients giving their consent for the study
* Body mass index between 28 and 35 kg/m2 with co-morbid condition (type 2 diabetes, hypertension, dyslipidemia, obstructive sleep apnea, non-alcoholic fatty liver disease or invalidating joint pain)
* No weigh loss following life-style changes

Exclusion Criteria:

* Antibiotic treatment during the three previous months
* Patients at risk of gastric cancer requiring regular endoscopic surveillance
* Gastric localization of Crohn disease
* Portal hypertension
* Severe hepatic or renal failure
* Ongoing peptic ulcer
* Severe associated disease
* History of previous bariatric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate obesity undergoing endoscopic sleeve gastroplasty
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Serum metabolite profile using widely targeted metabolomics according to weigh loss amount (less than 10% of total weight versus more than 10% of total weight loss at 12 months post-surgery) | Before endoscopic sleeve gastroplasty
  A volume of 50 µl of serum/plasma will be used for analysis of serum metabolites using widely targeted metabolomics mass spectrometry.

SECONDARY OUTCOMES:
Clinical parameters at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  Weight expressed in kg, percentage of total weight loss and percentage of excessed weight loss will be analysed as they are systematically available in usual clinical practice.
Basic serum lipid profile at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  Basic serum lipid profile will be analysed by spectrometry as they are systematically available in usual clinical practice.
Glycated hemoglobin at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  Glycated hemoglobin expressed in % will be analysed as they are systematically available in usual clinical practice.
Insulin at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  Insulin expressed in mUI/l will be analysed as it is systematically available in usual clinical practice.
C peptide at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  C peptide expressed in µg/l will be analysed as it is systematically available in usual clinical practice.
Ferritin at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  Ferritin expressed in µg/l will be analysed as it is systematically available in usual clinical practice.
Liver function test parameter Alanine transaminase (ALT) at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  ALT levels expressed in IU/l will be analysed as they are systematically available in usual clinical practice.
Liver function test parameter aspartate transaminase (AST) at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  AST levels expressed in IU/l will be analysed as they are systematically available in usual clinical practice.
Liver function test parameter Gamma-glutamyltransferase (GGT) at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  GGT levels expressed in IU/l will be analysed as they are systematically available in usual clinical practice.
Liver function test parameter Alkaline phosphatase (ALP) at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  ALP levels expressed in IU/l will be analysed as they are systematically available in usual clinical practice.
Liver fibrosis assessed by transient elastometry at baseline and then at 3 and 12 month post-intervention | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  Transient elastometry expressed in kPa will be analysed as they are systematically available in usual clinical practice.
Liver steatosis assessed by controlled attenuation parameter (CAP) at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  Controlled attenuation parameter expressed in dB/m will be analysed as they are systematically available in usual clinical practice.
Serum metabolites using widely targeted metabolomics at baseline and then at 3 and 12 month post-intervention. | Change from baseline (before endoscopic sleeve gastroplasty) to Month 3 and Month 12
  A volume of 50 µl of serum/plasma will be used for analysis of serum metabolites using widely targeted metabolomics by mass spectrometry.
Complications of endoscopic sleeve gastroplasty | During the first week post-endoscopic sleeve gastroplasty and at Month 3 and Month 12
  Data on the potential complications (occurrence of perforation, bleeding, peritonitis and other infections, thrombo-embolic events and death) of endoscopic sleeve gastroplasty will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Cosmin VOICAN, MD, PhD, Principal Investigator — APHP, Antoine-Béclère Hospital